CLINICAL TRIAL: NCT02938429
Title: Physical Activity Measured Through Accelerometers and Its Association With Endothelial Function in Young Patients With Fontan Physiology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Pro00060485
Record Dates: First submitted 2016-10-17; First posted 2016-10-19 (Estimated); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Heart Defects
Keywords: congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Participants with Fontan circulation (Other): Physical activity measurements: Participants will wear Actigraph GT3X+ accelerometers for 7 consecutive days and complete a physical activity log. Data from the accelerometers and physical activity log will be cross referenced.
  Endothelial function measurements: Participants undergo Digital Thermal Monitoring (DTM) via Vendys (VENDYS-6000, Endothelix Inc., Houston, TX). Since DTM is not currently a validated tool and its use has not been published in a paediatric population, we will employ a second assessment of endothelial function, the Endothelial Pulse Amplitude Test (Endo-PAT, Itamar Medical).
  Participants will complete a questionnaire to access factors that can affect endothelial function.
  Interventions: Other: Physical activity measures via Actigraph GT3X+ accelerometers for 7 consecutive days
- Age and gender matched controlled (Other): Physical activity measurements: Participants will wear Actigraph GT3X+ accelerometers for 7 consecutive days and complete a physical activity log. Data from the accelerometers and physical activity log will be cross referenced.
  Endothelial function measurements: Participants undergo Digital Thermal Monitoring (DTM) via Vendys (VENDYS-6000, Endothelix Inc., Houston, TX). Since DTM is not currently a validated tool and its use has not been published in a paediatric population, we will employ a second assessment of endothelial function, the Endothelial Pulse Amplitude Test (Endo-PAT, Itamar Medical).
  Participants will complete a questionnaire to access factors that can affect endothelial function.
  Interventions: Other: Physical activity measures via Actigraph GT3X+ accelerometers for 7 consecutive days

INTERVENTIONS:
Other: Physical activity measures via Actigraph GT3X+ accelerometers for 7 consecutive days
  Other Names: Endothelial function measurements: Digital Thermal Monitoring (DTM) via Vendys (VENDYS-6000, Endothelix Inc., Houston, TX); Endothelial function measurements: Endothelial Pulse Amplitude Test (Endo-PAT, Itamar Medical)

SUMMARY:
This study will be a cross sectional assessment of physical activity as measured through accelerometers and its association with endothelial function of children with Fontan circulation and healthy age and gender matched controls who are followed at the University of Alberta - Stollery Children's hospital.

ELIGIBILITY:
Inclusion Criteria:

1. Children with Fontan physiology between the ages 24 months to 18 years at the Stollery Children's Hospital
2. Informed written consent obtained prior to enrolment
3. At least 6 months post Fontan procedure

Exclusion Criteria:

1. Patient hospitalized within the previous 2 weeks
2. Patient unable to ambulate independently
3. Underwent coarctation of the aorta repair using a subclavian flap.

Ages: 24 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Physical activity measured by accelerometers | Once consent/assent is obtained, participants will be asked to wear an Actigraph GT3X+ accelerometers for seven consecutive days, during waking hours.
Endothelial function measured by Digital Thermal Monitoring (DTM) via the automated, operator-independent protocol (VENDYS-6000, Endothelix Inc., Houston, TX) and the Endothelial Pulse Amplitude Test (Endo-PAT, Itamar Medical). | Once consent/assent is obtained, endothelial function will be measured one time during a routine clinical visit.

SECONDARY OUTCOMES:
Vascular health questionnaire | Once during routine clinical visit after informed consent/assent.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Conway, MD, Principal Investigator — University of Alberta
Locations (1):
- Stollery Children's Hospital, Edmonton, Alberta, Canada